CLINICAL TRIAL: NCT04184817
Title: Retrospective Clinical Study to Evaluate of Cranio-vertebral Abnormalities Through Radiological Analysis in Patients With Achondroplasia Treated/Followed at the Hôpital Femme Mère Enfant
Brief Title: Radiological Analysis on Patients With Achondroplasia Disorder
Acronym: Achondroplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: Achondroplasia_2019
Record Dates: First submitted 2019-11-25; First posted 2019-12-04 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2019-11

CONDITIONS: Achondroplasia
Keywords: Achondroplasia; cranio-vertebral abnormalities
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical data collection: The medical data of patients diagnosed by Achondroplasia will be collected. The radiological data will analyse to evaluate the severity of stenosis as well as its clinical tolerance and evolution.
  Interventions: Other: Collection of clinical data registered in Easily software

INTERVENTIONS:
Other: Collection of clinical data registered in Easily software — Collection of clinical data registered in Easily software

SUMMARY:
Achondroplasia is a genetic disorder characterized by disproportionate short stature. It affects about 1 in 2500 live births in the world. The cause of Achondroplasia was identified to be a gain-of-function mutations in the fibroblast growth receptor 3 (FGFR3). In these children compression of the spinal cord at the foramen magnum stenosis can occur in early childhood which, can lead to central sleep apnea. It can lead to morbidity and mortality. A surgical intervention may be indicated in patients who present a foramen magnum stenosis. However, surgical indications are still under discussion. The objective of this retrospective study is to analyse the degree of stenosis and its clinical tolerance/evolution from radiological data monitored at the Hospital Femme Mère Enfant.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls.
* Aged from 0 to 18 years old.
* Subjects with an Achondroplasia diagnosis.
* Patients or parents/ legal guardian must provide non opposition prior to participation in the study.

Exclusion Criteria:

- Patients or patient's parents or legal guardian whose have an objection for using their data.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Achondroplasia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the degree of foramen magnum stenosis, its clinical tolerance and its evolution by radiological clinical data of the patients with Achondroplasia | MRI results in children with Achondroplasia will be collected through study completion an average of 2 year.
  All patients with Achondroplasia pathology followed at the Hôpital Femme Mère Enfant can be included in this study. The patients can present spinal column abnormalities such as foramen magnum stenosis. All patients diagnosed with Achondroplasia had the MRI. The MRI results will be used to evaluate the degree of deformity of stenosis and its clinical tolerance as well as its evolution. These results will help us to detect the compression at the foramen magnum to prevent lethal complications.
  The endpoint choice of this retrospective study will be the MRI of the first visit and the last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Federico DI ROCCO, Pr, Principal Investigator — Hospices Civils de Lyon; Massimiliano Rossi, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme-Mère-Enfant, Bron, France